CLINICAL TRIAL: NCT05388981
Title: A Randomized, Placebo-Controlled Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of SBT115301 in Healthy Participants
Brief Title: Study of Single Doses of SBT115301 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sonoma Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBT115301-01
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-09

CONDITIONS: Safety
Keywords: healthy volunteers; safety

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, sequential escalating dose cohorts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Experimental): Intramuscular (IM) dose level 1
  Interventions: Biological: SBT115301; Biological: Placebo
- Cohort 2 (Experimental): IM dose level 2
  Interventions: Biological: SBT115301; Biological: Placebo
- Cohort 3 (Experimental): IM dose level 3
  Interventions: Biological: SBT115301; Biological: Placebo
- Cohort 4 (Experimental): IM dose level 4
  Interventions: Biological: SBT115301; Biological: Placebo
- Cohort 5 (Experimental): Intravenous (IV) dose level 1
  Interventions: Biological: SBT115301; Biological: Placebo

INTERVENTIONS:
Biological: SBT115301 — Immunomodulatory dimeric fusion protein
Biological: Placebo — Matched placebo

SUMMARY:
This study will test the safety and effects of SBT115301 when given as a single dose to healthy adult volunteers. It is the first study being done in humans. Increasing dose levels will be given after the safety at lower dose levels is shown. Some participants will receive placebo, and neither the participants or the study staff will know what drug (SBT115301 or placebo) is being given.

ELIGIBILITY:
Inclusion Criteria:

* Males or females not of childbearing potential
* Healthy participants based on medical history, physical examination, vital signs, electrocardiogram, and clinical laboratory tests
* Use of highly effective methods of contraception (sexually active males with partners of childbearing potential)
* Up-to-date vaccinations for coronavirus disease (COVID-19) and influenza

Exclusion Criteria:

* Chronic or acute illness
* History of drug or alcohol abuse or positive drug or alcohol screening results
* Clinically significant ECG abnormality
* Received attenuated live vaccine within 1 month or COVID-19 vaccine within 2 weeks prior to study, or anticipated vaccination during study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Adverse events | Day of treatment to end of follow-up period (71 days for Cohorts 1-4; 140 days for Cohort 5)
  Number of participants with treatment-emergent adverse events
Serious adverse events | Baseline to end of follow-up period (71 days for Cohorts 1-4; 140 days for Cohort 5)
  Number of participants with serious adverse events

SECONDARY OUTCOMES:
SBT115301 Serum Concentration | Day 1 to Day 72 (Cohorts 1-4) or Day 141 (Cohort 5)
  Serum concentration of SBT115301
Pharmacokinetic Parameters: Cmax | Day 1 to Day 72 (Cohorts 1-4) or Day 141 (Cohort 5)
  Maximum serum concentration (Cmax) of SBT115301
Pharmacokinetic Parameters: Tmax | Day 1 to Day 72 (Cohorts 1-4) or Day 141 (Cohort 5)
  Time of maximum SBT115301 serum concentration (Tmax)
Pharmacokinetic Parameters: AUC(0-last) | Day 1 to Day 72 (Cohorts 1-4) or Day 141 (Cohort 5)
  Area under the serum concentration-time curve (AUC) from time 0 to the last measurable serum concentration
Pharmacokinetic Parameters: AUC(0-inf) | Day 1 to Day 72 (Cohorts 1-4) or Day 141 (Cohort 5)
  Area under the serum concentration-time curve from time 0 extrapolated to infinity
Pharmacokinetic Parameters: t1/2 | Day 1 to Day 72 (Cohorts 1-4) or Day 141 (Cohort 5)
  Terminal elimination half-life (t1/2)
Anti-Drug Antibodies | Day 1 to Day 72 (Cohorts 1-4) or Day 141 (Cohort 5)
  Number of participants with anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Valentine, DO, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No